CLINICAL TRIAL: NCT04660305
Title: Phase 1 Single Dose, Randomised, Double-blind, Two-way Crossover, Glucose Clamp Study Investigating the Pharmacodynamics, Pharmacokinetics and Safety of Arecor Rapid-acting Concentrated Insulin Aspart (AT278) in Comparison to Insulin Aspart NovoRapid® in Participants With Type 1 Diabetes Mellitus (T1DM).
Brief Title: AT278 and NovoRapid® in Glucose Clamp Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arecor Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARE-278-102
Record Dates: First submitted 2020-12-03; First posted 2020-12-09 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2020-12

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AT278 (Experimental): Single subcutaneous injection 0.3U/kg
  Interventions: Drug: AT278; Drug: NovoRapid
- NovoRapid (Active Comparator): Single subcutaneous injection 0.3U/kg
  Interventions: Drug: AT278; Drug: NovoRapid

INTERVENTIONS:
Drug: AT278 — Concentrated rapid acting insulin aspart
Drug: NovoRapid — Rapid acting insulin aspart
  Other Names: NovoLog

SUMMARY:
A phase 1, randomised, single-centre, double-blind, single-dose, two period balanced cross over study in a glucose clamp setting. The study compares the pharmacodynamic, pharmacokinetic and safety characteristics of AT278 and NovoRapid® in male participants with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of type 1 diabetes for at least 12 months
2. Receiving treatment with multiple daily insulin injections or insulin pump therapy for at least 12 months
3. HbA1c concentration ≤8.5% at screening
4. Weight within the range 75kg - 100kg (both inclusive)

Exclusion Criteria:

1. Known or suspected hypersensitivity to Investigational Medicinal Products
2. Clinically significant concomitant disease or abnormal lab values
3. Supine systolic BP outside range 95-140mmHg and/or diastolic BP greater than 90mmHG

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2021-06-03 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
Area under the glucose infusion-rate curve of insulin aspart | 0 - 8 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trials Unit, Medical University of Graz, Graz, Austria